CLINICAL TRIAL: NCT06974032
Title: Expanding the Use of Paracervical Block for IUD Placements and Adding a Compassionate Care Assessment- Aim 3
Brief Title: Empathy Through Pain Control: Lidocaine Gel vs. Placebo Prior to IUD Placement
Acronym: EPIC3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 812588
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Contraception; Pain, Acute; Anesthesia, Local
MeSH Terms: conditions — Acute Pain | interventions — phenylmercury borate

STUDY DESIGN:
Intervention Model Description: Two-armed double-blind, randomized controlled
Who Masked: Participant, Care Provider
Masking Description: Participants will not know their group assignment. Clinicians will not know which group the participant is in. The gel will be prepared by another member of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% lidocaine gel (Xylocaine) (Experimental): Experimental group: will receive 6cc of 2 lidocaine gel (Xylocaine) administered vaginally before paracervical block for IUD placement
  Interventions: Drug: Xylocaine jelly 2%
- Non-Medicated Gel (Surgilube) (Placebo Comparator): Placebo group: will receive 6cc of non-medicated (surgilube) gel administered vaginally before paracervical block for IUD placement
  Interventions: Drug: Surgilube

INTERVENTIONS:
Drug: Xylocaine jelly 2% — To determine if a 6cc of 2% lidocaine jelly decreases pain of paracervical block injection before IUD placement in nulliparous women
  Arms: 2% lidocaine gel (Xylocaine)
Drug: Surgilube — To determine if the placebo gel increases pain of paracervical block injection before IUD placement in nulliparous women
  Arms: Non-Medicated Gel (Surgilube)

SUMMARY:
The goal of this research study is to learn more about how different uses of a numbing medication might affect pain levels while getting an IUD placed. The investigators are also studying patients' opinions of their clinicians' empathy.

The investigators are inviting patients who have never given birth who arrive at their clinic visit seeking an IUD.

Usually, at University of California, San Diego (UCSD), for patients who have never delivered, clinicians numb both the sides of the cervix with a lidocaine-based paracervical block. The purpose of this research study is to compare perceptions of pain between lidocaine-infused gel and non-medicated gel inserted into the vagina before paracervical block and IUD placement for nulliparous women.

DETAILED DESCRIPTION:
Lidocaine Jelly is a substance that has been approved by the Food and Drug Administration (FDA). At UCSD and other places, it is not currently standard practice for people with prior deliveries birth to receive any sort of vaginal jelly before paracervical block prior to IUD placement.

Participants who take part in this study, may receive 6cc of 2% lidocaine gel or 6cc of a non-medicated gel in the vagina before a paracervical block for IUD placement.

Throughout the local anesthetic and intrauterine device (IUD) placement procedure, research team members will present participants with questionnaires to complete to assess participants' pain, participants' satisfaction with the procedure, and how much empathy participants feel the clinician has shown.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Women presenting for IUD placement for contraception or heavy menstrual bleeding
3. Ages 18-50
4. English-speaking
5. Participants must not have a past medical history of substance use disorders, pain disorders, use of prescription pain medications or are found to be pregnant
6. Nulliparous (never given birth)

Exclusion Criteria:

1. History of ever giving birth
2. Current use of prescription pain medication prior to procedure. Over-the-counter medications such as those containing ibuprofen, aspirin, acetaminophen, or naproxen are allowed.
3. Diagnosed chronic pain condition
4. Current pregnancy
5. Known allergic reactions to components of the local anesthetic
6. History of an IUD placement
7. Current substance use or history of substance use
8. Known contraindications to IUD, such as unexplained vaginal bleeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain scores during IUD placement procedure | From speculum placement to 5 minutes post-procedure
  Does 2% lidocaine jelly decrease pain of paracervical block injection before IUD placement procedures among nulliparous women? Pain will be measured on a 10-cm Visual Analog Scale (VAS) with score points ranging from 0-10, where 0 means "No pain" and 10 means "Worst pain possible."
Patient perceptions of clinician empathy | From pre-procedure baseline to 5 minutes post-procedure
  What is the relationship between pain and feelings about clinician empathy? Empathy will be measured through answers to the 10-question Consultation and Relational Empathy (CARE) Measure. Each question is answered by a 5-point scale of how well the patient believes their clinician to be at various types of empathetic gestures, where 1 equals "poor" and 5 equals "excellent."

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K Mody, MD, MPH, Principal Investigator — UC San Diego

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin J, Kaneshiro B, Elia J, Raidoo S, Savala M, Soon R. Buffered lidocaine for paracervical blocks in first-trimester abortions: a randomized controlled trial. Contracept X. 2020 Oct 18;2:100044. doi: 10.1016/j.conx.2020.100044. eCollection 2020. PMID 33196038
- [Background] Azizkhani R, Forghani M, Maghami-Mehr A, Masomi B. The effects of injections of warmed bicarbonate-buffered Lidocaine as a painkiller for patients with trauma. J Inj Violence Res. 2015 Jul;7(2):87-8. doi: 10.5249/jivr.v7i2.523. Epub 2013 Dec 12. No abstract available. PMID 24879075
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Welch MN, Czyz CN, Kalwerisky K, Holck DE, Mihora LD. Double-blind, bilateral pain comparison with simultaneous injection of 2% lidocaine versus buffered 2% lidocaine for periocular anesthesia. Ophthalmology. 2012 Oct;119(10):2048-52. doi: 10.1016/j.ophtha.2012.05.029. Epub 2012 Jul 6. PMID 22771049
- [Background] Narvaez J, Wessels I, Bacon G, Chin VR, Baqai WK, Zimmerman GJ. Prospective randomized evaluation of short-term complications when using buffered or unbuffered lidocaine 1% with epinephrine for blepharoplasty surgery. Ophthalmic Plast Reconstr Surg. 2010 Jan-Feb;26(1):33-5. doi: 10.1097/IOP.0b013e3181b80c13. PMID 20090482
- [Background] Hobeich P, Simon S, Schneiderman E, He J. A prospective, randomized, double-blind comparison of the injection pain and anesthetic onset of 2% lidocaine with 1:100,000 epinephrine buffered with 5% and 10% sodium bicarbonate in maxillary infiltrations. J Endod. 2013 May;39(5):597-9. doi: 10.1016/j.joen.2013.01.008. Epub 2013 Mar 20. PMID 23611375
- [Background] Harreld TK, Fowler S, Drum M, Reader A, Nusstein J, Beck M. Efficacy of a Buffered 4% Lidocaine Formulation for Incision and Drainage: A Prospective, Randomized, Double-blind Study. J Endod. 2015 Oct;41(10):1583-8. doi: 10.1016/j.joen.2015.06.017. Epub 2015 Aug 4. PMID 26253800
- [Background] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115
- [Background] Allen RH, Raker C, Goyal V. Higher dose cervical 2% lidocaine gel for IUD insertion: a randomized controlled trial. Contraception. 2013 Dec;88(6):730-6. doi: 10.1016/j.contraception.2013.07.009. Epub 2013 Aug 1. PMID 24012096